CLINICAL TRIAL: NCT02821975
Title: Evaluating Cognitive Computer Training as a Tool for Returning Earlier to Work After Depression
Brief Title: Cognitive Computer Training in Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cognex-depression
Record Dates: First submitted 2016-06-06; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Depression in Remission; Cognitive Computer Training; Returning to Work
Keywords: Depression; Cognitive function; Work
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive computer training (Experimental): This is the intervention group receiving cognitive computer training three times a week for three months.
  Interventions: Other: Cognitive computer training
- cogntrol group (No Intervention): The control group do not receive cognitive computer training for three months

INTERVENTIONS:
Other: Cognitive computer training — COGNIFIT is cognitive computer training. Its purpose is to improve cognitive function and is designed to accommodate each individual's cognitive strengths and weaknesses. The cognitive computer training last three months and must be done three times a week, in session lasting 10-20 minutes.
  Other Names: Cognifit personalized training
  Arms: Cognitive computer training

SUMMARY:
Cognitive impairment plays an important role in functional recovery and leads to long-term sickness absence. Therefore there is a need of a treatment specifically improving cognitive functions. In this pilot study the investigators aim to evaluate the feasibility of using cognitive computer training in patients with unipolar depression to enhance cognitive performance. Further the investigators investigate whether this intervention shortens sick leave.

DETAILED DESCRIPTION:
This study will evaluate cognitive computer training on patients in remission from depression by measuring the compliance and effect, investigating whether patients returned earlier to work and examine patients' physical and psychological health. This is done by comparing an intervention group and a control group.

Outpatients from psychiatric department Odense in Denmark will be recruited from December 2015 to July 2017.

At enrolment the participants wil be randomized 1:1 to either the intervention group or the control group. After the participants will complete a clinical interview and answer the The Short Form (36) Health Survey (SF-36) questionnaire. The participants' cognitive function and depression severity will be measured at baseline and three months follow-up. At nine months follow-up the participants will receive an email with the SF-36 questionnaire and questions about their education and work status, which they were required to answer.

The intervention is a cognitive computer program, consisting of different computer games. The intervention will start at enrolment and finish at the three months follow-up. The participants in the intervention group will do trainings session lasting 10-20 minutes three times a week. Each participant ends up with a total of 36 training sessions.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of a moderate to severe unipolar depression according to the International Classification of Diseases -10 criteria
* receiving antidepressant medicine
* completed their treatment for depression
* not be in any risk of suicide
* study or work on reduced hours, be unemployed or on long-term sickness leave at enrolment.

Exclusion Criteria:

* neurological disease of the central nervous system
* alcohol or substance abuse
* pregnancy
* receiving disability pension
* receiving electroconvulsive therapy within the last 6 weeks.

Ages: 20 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Employment status of the participants at nine months follow-up | When the study is completed, approximately 15 months
  Questionnaire about employment status and will be send to the participants via email at nine months follow-up. The questionnaire include questions according to: current working situation; why they are not working; when they started working; do they work at the same workplace; do they have the same work assignments as before they got ill; do whey work the same number of hour as before the got ill.

SECONDARY OUTCOMES:
The difference in concentration from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Concentration is measured by The Digit Span Test
The difference in attention from baseline to 3 months follow-up in the intervention group compared to the control group | approximately nine months
  Attention is measured by The Letter Cancellation Test
The difference in working memory from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Working memory is measured by The Letter Number Sequencing
The difference in learning from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Learning is measured by the Rey Auditory Verbal Learning Test.
The difference in executive function from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Executive function is measured by The Verbal Fluency
The difference in psychomotor speed from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Psychomotor speed is measured by The Trial Making Test (TMT).
The difference in executive function from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  Executive function is measured by The Tower of London

OTHER OUTCOMES:
Compliance of cognitive computer training | approximately nine months
  The participants were supposed to do 36 sessions of cognitive computer training during three months. The actual completed trainings sessions are available on the website of the cognitive computer training, called COGNIFIT. The compliance is defined as the percentage of actual completed training sessions of the 36 sessions of training.
The difference in health status from baseline to 9 months follow-up in the intervention group compared to the control group. | approximately 15 months
  The health status is measured by a patient-reported survey called the The Short Form (36) Health Survey (SF-36) questionnaire
The difference in depression severity from baseline to 3 months follow-up in the intervention group compared to the control group. | approximately nine months
  The depression severity is measured by Hamilton Rating Scale for Depression (17-items)

CONTACTS AND LOCATIONS:
Overall Officials: Bent Nielsen, Prof.MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Research Unit of Psychiatry, Psychiatric Unit Odense - University function, Odense C, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No